CLINICAL TRIAL: NCT06278987
Title: Comparison of Cryoablation of Pericapsular Nerve Group (PENG) to Fascia Iliaca Catheter in Patients With a Hip Fracture
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANES-2024-32661
Record Dates: First submitted 2024-01-30; First posted 2024-02-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hip Fractures
Keywords: Hip fractures
MeSH Terms: conditions — Hip Fractures | interventions — Cryosurgery

STUDY DESIGN:
Intervention Model Description: This is a randomized prospective controlled trial. This will be single blinded trial. Randomization will be 1:1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG block and cryoablation (Experimental): Patients undergoing hip fracture repair aged 18-85
  Interventions: Drug: PENG block and cryoablation
- fascia iliaca compartment block (Experimental): Patients undergoing hip fracture repair aged 18-85
  Interventions: Drug: fascia iliaca compartment block

INTERVENTIONS:
Drug: PENG block and cryoablation — will receive an ultrasound guided PENG block with 20 mL of 0.5% bupivacaine followed by cryoablation of the PENG nerves.
  Arms: PENG block and cryoablation
Drug: fascia iliaca compartment block — will receive an ultrasound guided fascia iliaca compartment catheter with initial bolus of 20 mL of 0.5% bupivacaine followed by infusion of 0.2% ropivacaine at 10 mL per hour
  Arms: fascia iliaca compartment block

SUMMARY:
The purpose of this study is to determine if patients with hip fractures who undergo cryoablation of the PENG have improved pain control 30 days from surgery when compared to those who have a fascia iliaca catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip fracture repair aged 18-85.

Exclusion Criteria:

* Patients who have an exclusion to regional anesthesia.
* Patients who are pregnant assessed via self-report or pregnancy test if they have taken one.
* Non-English speakers
* Patients who already had their fracture repaired"

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximum pain score on Post-operative day 30 | 30 days post surgery
  Maximum pain score on day 30 post surgery. Pain Scale is 0-10 with 0 meaning no pain (better outcome) and 10 meaning worst pain imaginable (worse outcome).
Opioid use | day 0, 1, 2, 3, 4, 5, 6, 7 post surgery
  Opioid use and Functional Pain scores on POD 0, 1, 2, 3, 4, 5, 6, 7 - measured in milligrams morphine equivalents
functional pain scores | day 0, 1, 2, 3, 4, 5, 6, 7 post surgery post surgery
  Functional Pain Score on Post Operative Day 0, 1, 2, 3, 4, 5, 6, 7 - measured with Pain Scale 0-10 with 0 meaning no pain (better outcome) and 10 meaning worst pain imaginable (worse outcome)
number of patients using opioids | 30 days post surgery
  measured in number of patients
Length of Hospital Stay | 30 days post surgery
  measured in number of days
Time to first ambulation | 30 days post surgery
  measured in Days:Hours:Minutes post operation
Number of patients returned home by Post Operative Day 30 | 30 days post surgery
  measured in number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Jason Habeck, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States